CLINICAL TRIAL: NCT00184314
Title: Follow-up Eating Disorder Patients and Their Parents Leaving Treatment From 1988 to 2002 at Child and Adolescent Department at Levanger Hospital.
Brief Title: Follow-up of Eating Disorder Patients From a 15-year Period.
Status: Completed | Type: Observational
Sponsor: Norwegian University of Science and Technology (Other)
Collaborators: Helse Nord-Trøndelag HF (Other)
Responsible Party: Sponsor
Other Study IDs: 148-02
Record Dates: First submitted 2005-09-13; First posted 2005-09-16 (Estimated); Last update posted 2017-02-09 (Estimated); Status verified 2017-02

CONDITIONS: Eating Disorder Symptoms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Retrospective follow-up study of former eating disorder patients in child- and adolescent psychiatry on psychiatric symptoms and social intelligence.

DETAILED DESCRIPTION:
Former patients and their parents were contacted 3 to 15 years after their completed treatment for eating disorders at Levanger Hospital, Child and Adolescent Psychiatry Department, in the period from 1988 to 2002. Interviews focusing on general psychiatric symptom, specific eating disorder symptoms, social intelligence and consumer satisfaction. Parents were also contacted and interviewed on consumer satisfaction.

ELIGIBILITY:
Inclusion Criteria:

* Eating disorder symptoms or disorder

Exclusion Criteria:

-

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: former eating disorder patients
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2004-03 (Actual); Primary Completion 2004-08 (Actual); Study Completion 2004-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tormod Rimehaug, ass.prof., Principal Investigator — Norwegian University of Science and Technology (NTNU), Faculty of Medicine, Dep of Neuroscience, Center For Child And Adolescent Mental Health
Locations (1):
- Child Psychiatry Department, Levanger Hospital, Levanger, Levanger, Norway

REFERENCES:
- [Result] Wanderås C. Do Individuals with Eating Disorders Have Lower Emotional Intelligence?: Are Eating Disorders Comorbid with Low Emotional Intelligence? Doctoral dissertation, Institute of Psychology, Aarhus University, 2005